CLINICAL TRIAL: NCT06071325
Title: Green Digital Diabetes Waste Project: Quantifying the Amount of Environmental Waste Associated With Devices and Technology
Brief Title: Green Digital Diabetes Waste Project
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Collaborators: Diabetes Technology Society (Other)
Responsible Party: Principal Investigator, Jing Wang, Principal Investigator, Florida State University
Other Study IDs: STUDY00004453
Record Dates: First submitted 2023-10-03; First posted 2023-10-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: Continuous glucose monitor; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus; Multiple daily injection; Insulin pump; Diabetes waste
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AID Group: We anticipate enrolling between 30 and 50 participants who will be recruited to participate in the Automated Insulin Delivery (AID) system study.
- MDI + CGM Group: We anticipate that between 10 and 30 participants will be enrolled in the study and will be utilizing Multiple Daily Injections (MDI) therapy in conjunction with Continuous Glucose Monitoring (CGM). MDI therapy will be defined as administering three or more injections per day.

SUMMARY:
The purpose of this study is to determine how people with diabetes are disposing of various products and devices and at what rates so that better devices with less waste can be designed in the future.

DETAILED DESCRIPTION:
The study aims to compare the amount of environmental waste that is generated during the management of diabetes of participants who are using a CGM and on multiple daily injection (MDI) or using an AID (automated insulin delivery) system. This study is expected to demonstrate which devices create the most waste and where opportunities exist to decrease diabetes device waste. We will collect data to describe both quantitatively (via daily survey) and qualitatively (via photography) the types of waste that are generated during the management of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Person with diabetes (self-identified), either type 1 or type 2, who has been diagnosed at least 6 months earlier
* Age 18 years and above
* Use of a CGM
* Use of an insulin pump or on MDI
* Access to the Internet and e-mail
* Access to a smartphone with photographic capability
* Able and willing to provide informed consent

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Any condition which, in the opinion of an investigator, would make the subject not qualified to participate in the study.
* Adults unable to consent
* Adults unable to speak English
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Cognitively impaired adults

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosed diabetes mellitus (either Type 1 or Type 2) at least 6 months earlier, and treated with insulin and a continuous glucose monitor (CGM).
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Types and Amount of Diabetes Waste | 30 days
  Types and Amount of Environmental Waste Related to Diabetes Management as Measured Quantitately by Survey and Qualitatively by Photos

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PhD, Principal Investigator — Dean & Prof. of FSU College of Nursing; David C Klonoff, MD, Principal Investigator — President of Diabetes Technology Society and Clinical Professor of UCSF Medicine
Locations (2):
- United States (2):
  - Diabetes Technology Society, Burlingame, California
  - Florida State University, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers